CLINICAL TRIAL: NCT00002526
Title: Continuous 5 Days Infusion of High Dose Ifosfamide and Adriamycin in Patients With Advanced Sarcoma
Brief Title: Chemotherapy in Treating Patients With Advanced Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 57/93; EU-93004
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Ovarian Cancer; Sarcoma
Keywords: stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; ovarian sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Ovarian Neoplasms; Sarcoma | interventions — Filgrastim; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: doxorubicin hydrochloride
Drug: ifosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of ifosfamide and doxorubicin in patients with advanced sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, time to treatment failure, and survival in patients with advanced soft tissue or gynecological sarcoma treated with high-dose ifosfamide and doxorubicin.

OUTLINE: Patients receive ifosfamide IV continuously on days 1-5 and doxorubicin IV on days 1-3. Filgrastim (G-CSF) is administered subcutaneously daily beginning 24 hours after completion of ifosfamide infusion and continuing through day 16 (or until day 20 if blood counts have not recovered by day 16). Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed at treatment failure and then annually thereafter.

PROJECTED ACCRUAL: A total of 16-46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced soft tissue or gynecologic sarcoma Measurable disease No brain metastases (CT scan required if metastases are clinically suspected)

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: WHO 0-2 Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Liver function tests no greater than 2 times normal Albumin 4.0-6.0 g/dL Renal: Creatinine clearance at least 60 mL/min Cardiovascular: Cardiac function normal by MUGA scan or echocardiogram Other: No other prior or concurrent malignancy except radically removed nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the bladder No prior radiotherapy to indicator lesion Surgery: Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1993-01; Primary Completion 1995-09 (Actual); Study Completion 1995-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Leyvraz, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Leyvraz S, Zweifel M, Jundt G, Lissoni A, Cerny T, Sessa C, Fey M, Dietrich D, Honegger HP; Swiss Group for Clinical Cancer Research. Long-term results of a multicenter SAKK trial on high-dose ifosfamide and doxorubicin in advanced or metastatic gynecologic sarcomas. Ann Oncol. 2006 Apr;17(4):646-51. doi: 10.1093/annonc/mdl020. Epub 2006 Feb 24. PMID 16500907